CLINICAL TRIAL: NCT01876927
Title: A Randomised Phase Ii Study Of Pre-Operative Or Peri-Operative Docetaxel, Oxaliplatin, Capecitabine (Dox) Regimen In Patients With Locally Advanced Resectable Gastric Cancer
Brief Title: Pre-Operative Or Peri-Operative Dox Regimen In Patients With Locally Advanced Resectable Gastric Cancer
Acronym: GastroDOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST151.01; 2010-020189-37 (EudraCT Number)
Record Dates: First submitted 2013-06-07; First posted 2013-06-13 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Gastric Cancer; Locally Advanced Malignant Neoplasm
Keywords: Locally; Advanced; Resectable; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): DOX 4 cycles - Surgery - Follow-up
  DOX:
  Docetaxel 35 mg/m2 day 1 and 8 by one hour infusion; Oxaliplatin 80 mg/m2 day 1 by two hours infusion; Capecitabine 750 mg/m2 x 2 daily for 2 weeks, per OS.
  Treatment should be administered for 4 cycles before surgery. Each cycle will be repeated every 3 weeks.
  Interventions: Other: DOX 4 cycles - Surgery
- Arm B (Experimental): DOX 2 cycles - Surgery - DOX 2 cycles - Follow-up
  DOX:
  Docetaxel 35 mg/m2 day 1 and 8 by one hour infusion; Oxaliplatin 80 mg/m2 day 1 by two hours infusion; Capecitabine 750 mg/m2 x 2 daily for 2 weeks, per OS.
  Treatment should be administered for 2 cycles before surgery and for further 2 cycles after surgery, unless progression of disease or unacceptable toxicity occurs, or patient refusal. In these cases patients will go off treatment.
  Each cycle will be repeated every 3 weeks.
  Interventions: Other: DOX 2 cycles - Surgery - DOX 2 cycles

INTERVENTIONS:
Other: DOX 4 cycles - Surgery — DOX 4 cycles - Surgery
  Arms: Arm A
Other: DOX 2 cycles - Surgery - DOX 2 cycles — DOX 2 cycles - Surgery - DOX 2 cycles
  Arms: Arm B

SUMMARY:
Study design:

Multicenter, randomized, open label phase II study Arm A: DOX 4 cycles - Surgery - Follow-up Arm B: DOX 2 cycles - Surgery - DOX 2 cycles - Follow-up

Population:

Male or female, 18-75 years of age, with a diagnosis of histologically confirmed, potentially resectable adenocarcinoma of the stomach.

Sample Size: Planned sample size is 90 patients, 45 patients for each arm (p0=50%, p1=80%, alpha=0.05 (two sides), beta=0.2)

Treatment Plan:

Treatment will be administered for 4 and 2 cycles before surgery in arm A and B, respectively, and in arm B for a further 2 cycles after surgery unless progression or unacceptable toxicity occurs, or a patient refuses treatment. In such cases patients will go off treatment. 3-6 weeks after the end of the fourth (arm A) or second (arm B) preoperative cycle, patients will undergo surgery.

After surgery 3-6 weeks from surgery patients in arm B will receive 2 more cycles.

DOX: Docetaxel 35 mg/m2 day 1 and 8 Oxaliplatin 80 mg/m2 day 1 Capecitabine 750 mg/m2 x 2 daily for 2 weeks

Cycles repeated every 3 weeks

Evaluation criteria: Tumor assessment will be performed according to the RECIST criteria (version 1.1).

Duration of Study:

Overall study duration: 07/2010- 03/2017 Planned study duration per patient: 5 years

DETAILED DESCRIPTION:
Title: A randomised phase II study of pre-operative or peri-operative docetaxel, oxaliplatin, capecitabine (DOX) regimen in patients with locally advanced resectable gastric cancer.

Clinical Phase: II

Study Objectives:

Primary:

The percentage of patients receiving all the planned chemotherapeutic cycles.

Secondary:

* Downstaging according to Recist criteria
* pT1-3 vs pT0.
* Safety: number of patients with grade 3-4 toxicity
* The role of PET Scan as predictor of response
* Curative vs palliative surgery
* TTP
* OS
* Diagnostic correlation between the various staging methods
* Possible correlations between CT scan, CT/PET, laparoscopy;
* Molecular markers related to toxicity: DPYD, MTHFR, TS, XPD, ERCC1, XRCC1;
* Molecular markers related to prognosis: TYMS, GSTP1, COX-2, RUNX3, methylation profile (Cox2, hMLH1, MGMT);
* Molecular markers related to therapy response: TYMS, DPYD, MTHFR, OPRT, ERCC1, XRCC1/2/3, GSTP1, GSTM1, GSTT1, ABCB1, methylation profile (Cox2, hMLH1, MGMT), whole genome arrayCGH.

Study design:

Multicenter, randomized, open label phase II study Arm A: DOX 4 cycles - Surgery - Follow-up Arm B: DOX 2 cycles - Surgery - DOX 2 cycles - Follow-up

Population:

Male or female, 18-75 years of age, with a diagnosis of histologically confirmed, potentially resectable adenocarcinoma of the stomach.

Sample Size: Planned sample size is 90 patients, 45 patients for each arm (p0=50%, p1=80%, alpha=0.05 (two sides), beta=0.2)

Treatment Plan:

Treatment will be administered for 4 and 2 cycles before surgery in arm A and B, respectively, and in arm B for a further 2 cycles after surgery unless progression or unacceptable toxicity occurs, or a patient refuses treatment. In such cases patients will go off treatment. 3-6 weeks after the end of the fourth (arm A) or second (arm B) preoperative cycle, patients will undergo surgery.

After surgery 3-6 weeks from surgery patients in arm B will receive 2 more cycles.

DOX: Docetaxel 35 mg/m2 day 1 and 8 Oxaliplatin 80 mg/m2 day 1 Capecitabine 750 mg/m2 x 2 daily for 2 weeks

Cycles repeated every 3 weeks

Evaluation criteria: Tumor assessment will be performed according to the RECIST criteria (version 1.1).

Duration of Study:

Overall study duration: 07/2010- 03/2017 Planned study duration per patient: 5 years

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consents
2. Male or female 18-75 years of age
3. Diagnosis of histologically confirmed, potentially resectable adenocarcinoma of the stomach
4. cT3 subserosal - cT4a - cT4b (7th edition UICC TNM) or bulky lymph node metastases independently of T
5. ECOG performance status of 0-1 at study entry
6. Laboratory requirements (≤ 7 days prior chemotherapy start):

   1. Hematology:

      I) Neutrophils > 1.5 x 109 /L II) Platelets > 100 x 109 /L III) Hemoglobin > 10g/dL
   2. Hepatic function I) Total bilirubin < 1.25 UNL II) AST (SGOT) and ALT (SGPT) < 2.5xUNL III) Alkaline phosphatase < 2.5xUNL
   3. Renal function I) Creatinine <1.5 UNL In the event of border-line values, the calculated creatinine clearance should be > 60 mL/min;

      * Written informed consent signed and dated before randomization procedures, including expected cooperation of patients for treatment and follow-up, must be obtained and documented according to local regulatory requirements.
      * Effective contraception for both male and female patients if the risk of conception exists

Exclusion Criteria:

1. Early gastric cancer (if N0)
2. T2 (according to 7th edition of UICC TNM) if N0
3. Linitis plastica
4. Positive peritoneal cytology
5. Distant metastases
6. Neoplasm involving the gastro-esophageal junction
7. Pertoneal involvement
8. Concurrent chronic systemic immune therapy
9. Any investigational agent(s) administered 4 weeks prior to entry
10. Clinically relevant coronary artery disease, a history of myocardial infarction or of hypertension not controlled by therapy within the last 12 months
11. Known grade 3 or 4 allergic reaction to any of the components of the treatment
12. Known drug abuse/alcohol abuse
13. Legal incapacity or limited legal capacity
14. Medical or psychological condition which, in the opinion of the investigator, would not permit the patient to complete the study or sign meaningful informed consent
15. Women who are pregnant or breastfeeding
16. Acute or subacute intestinal occlusion
17. Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for ≥ 5 years will be allowed to enter the trial)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2010-09; Primary Completion 2017-03 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
the difference in percentage of patients receiving all the planned chemotherapeutic cycles between the two arms. | 7 years

SECONDARY OUTCOMES:
The percentage of tumors downstaged at the diagnosis | 7 years
  To determine the percentage of tumors downstaged at the diagnosis, compared with the pathological stage detected at the time of surgery (according to Recist criteria)
Treatment tolerability and safety and tumor response in patients with pathological stage pT1-3 vs pT0 | 7 years
  Comparation of treatment tolerability and safety and tumor response between patients with pathological stage pT1-3 vs pT0 (detected at the time of surgery)
Number of patients with adverse events of grade 3-4 as a measure of safety and tolerability | 7 years
Diagnostic capability of PET | 7 years
  Evaluation of the role of PET as a tool to detect tumor response
Efficacy comparation between curative vs palliative surgery | 7 years
Time to progression | 7 years
Overall survival | 7 years
Diagnostic capability of CT scan, CT/PET and laparoscopy | 7 years
  Evaluation of possible correlations between the diagnostic techniques CT scan, CT/PET and laparoscopy
Biological profile of treatment toxicity | 7 years
  Biological detection of molecular markers related to treatment toxicity (DPYD, MTHFR, TS, XPD, ERCC1, XRCC1)
Biological profile of treatment prognosis | 7 years
  Biological detection of molecular markers related to treatment prognosis (TYMS, GSTP1, COX-2, RUNX3, methylation profile (Cox2, hMLH1, MGMT))
Biologcal profile of treatment response | 7 years
  Biological detection of molecular markers related to therapy response (TYMS, DPYD, MTHFR, OPRT, ERCC1, XRCC1/2/3, GSTP1, GSTM1, GSTT1, ABCB1, methylation profile (Cox2, hMLH1, MGMT), whole genome arrayCGH)

CONTACTS AND LOCATIONS:
Overall Officials: Manlio Monti, MD, Principal Investigator — IRST IRCCS, Meldola
Locations (20):
- Italy (20):
  - Azienda Ospedaliero - Universitaria Ospedali Riuniti Umberto I - GM Lancisi, Ancona, AN
  - USL 8 Arezzo - Presidio Ospedaliero Zona Casentino - Ospedale di Bibbiena, Bibbiena, AR
  - USL 8 Arezzo - Ospedale "Santa Maria alla Gruccia", Montevarchi, AR
  - UO Oncologia , Spedali Civili di Brescia, Brescia, BS
  - Ospedale Bufalini, Cesena, FC
  - UO oncologia medica IRCCS IRST, Meldola (FC), FC
  - UOC Oncologia , Azienda USL 11, Empoli, FI
  - Ospedale Careggi, Florence, FI
  - UO ONCOLOGIA , Istituto Europeo di Oncologia, Milan, MI
  - Istituto Clinico Humanitas, Rozzano, MI
  - Azienda Ospedaliera Universitaria Pisana, Pisa, PI
  - UO Oncologia, Fondazione Policlinico San Matteo, Pavia, PV
  - UO Oncologia Medica, PO Rimini, AUSL della Romagna, Rimini, RI
  - UO Oncologia , Casa di Cura Tortorella, Salerno, SA
  - Policlinico Le Scotte, Siena, SI
  - UO Oncologia, Azienda Ospedaliero Treviglio, Treviglio, TV
  - UO Oncologia Medica, azienda Ospedaliera di Varese, Varese, VA
  - Azienda Ospedaliera di Perugia - Ospedale S. Maria della Misericordia, Perugia
  - Ospedale San Filippo Neri, Roma
  - Ospedale Borgo Trento, Verona